CLINICAL TRIAL: NCT01310894
Title: A European Randomised Phase 3 Study to Assess the Efficacy and Safety of TOOKAD® Soluble for Localised Prostate Cancer Compared to Active Surveillance
Brief Title: Efficacy and Safety Study of TOOKAD® Soluble for Localised Prostate Cancer Compared to Active Surveillance.
Acronym: PCM301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1001 PCM301
Record Dates: First submitted 2011-03-01; First posted 2011-03-09 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostatic Disease; Genital Neoplasm,male; Urogenital neoplasm; Genital disease,male; Male urogenital disease; Neoplasms; Neoplasms by site; Prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Carcinoma | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TOOKAD® Soluble (Experimental): TOOKAD® Soluble, lyophilized formulation, given at a dose of 4mg/Kg.
  Interventions: Drug: TOOKAD® Soluble
- Active Surveillance (No Intervention): Active surveillance is one of the management strategy in men who have low-risk prostate cancer

INTERVENTIONS:
Drug: TOOKAD® Soluble — TOOKAD® Soluble-VTP procedure will consist of an IntraVenous (IV) administration to patients using a 753nm laser light at a fixed power of 150mW/cm and a fixed energy at 200J/cm delivered through transperineal interstitial optical fibers. The needles are positioned in the prostate under ultra sound image guidance
  Other Names: WST11
  Arms: TOOKAD® Soluble

SUMMARY:
The aims of this study are:

* to assess the impact of TOOKAD® Soluble-Vascular Targeted Photodynamic Therapy (VTP) on the rate of absence of definite cancer using patients on active surveillance as a comparison (co-primary objective A) and
* to determine the difference in rate of treatment failure associated with observed progression of disease from low risk prostate cancer to moderate or higher risk prostate cancer in men who undergo TOOKAD® Soluble-VTP compared to men on active surveillance (co-primary objective B).

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, open label, randomised controlled study in subjects diagnosed with low risk prostate cancer on TransRectal Ultrasound (TRUS) guided biopsy.

Subjects will be randomised to either Active Surveillance or TOOKAD® Soluble VTP. Subjects will remain in the study for approximately 24 months following randomisation. A total of 400 subjects will be entered into the study; 200 will receive Active Surveillance and 200 will receive TOOKAD® Soluble-VTP.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for inclusion in the study if all of the following criteria are met:

1. Low risk prostate cancer diagnosed using one transrectal ultrasound guided biopsy (TRUS)using from 10 to 24 cores performed less than 12 months prior to enrolment, and showing the following:

   * Gleason 3 + 3 prostate adenocarcinoma as a maximum,
   * Two (2) to three (3) cores positive for cancer
   * A maximum cancer core length of 5 mm in any core.
2. Cancer clinical stage up to T2a (pathological or radiological up to T2c disease permitted)
3. Serum prostate specific antigen (PSA) of 10 ng/mL or less
4. Prostate volume equal or greater than 25 cc and less than 70 cc.
5. Male subjects aged 18 years or older.

Exclusion Criteria:

Subjects will not be eligible for the study if meeting any of the following criteria:

1. Unwillingness to accept randomisation to either of the two arms of the study
2. Any prior or current treatment for prostate cancer, including surgery, radiation therapy (external or brachytherapy) or chemotherapy.
3. Any surgical intervention for benign prostatic hypertrophy
4. Life expectancy less than 10 years.
5. Any condition or history of illness or surgery that may pose an additional risk to men undergoing the VTP procedure.
6. Participation in another clinical study or recipient of an investigational product within 1 month of study entry.
7. Subject unable to understand the patient's information document, to give consent or complete the study tasks.
8. Subject in custody and or in residence in a nursing home or rehabilitation facility
9. Contra-indication to Magnetic resonance Imaging (MRI) (e.g., pacemaker, history of allergic reaction to gadolinium), or factors excluding accurate reading of pelvic MRI (e.g., hip prosthesis)
10. Any condition or history of illness or surgery that may pose an additional risk to men undergoing the TOOKAD® Soluble VTP procedure.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2011-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoint 'A': Rate of absence of definite cancer using patients on active surveillance as a comparison. | Month 24
  Histological changes are assessed using biopsies or any other pathology result obtained during the study planned or not.
Co-primary endpoint 'B': Difference in rate of treatment failure associated with observed progression of disease from low risk prostate cancer to moderate or higher risk prostate cancer. | Over 24 months follow-up.
  Moderate or higher risk is defined as the observation of:
  * More than 3 cores positive for cancer when considering all histological examination available during follow-up of study;
  * or any Gleason primary or secondary pattern 4 or more;
  * or at least one cancer core length greater than 5 mm;
  * or PSA>10ng/mL ( in 3 consecutive measures);
  * or any T3 prostate cancer,
  * or metastasis;
  * or prostate cancer related death

SECONDARY OUTCOMES:
The rate of additional prostate cancer radical therapy | Over 24 months follow-up
  Number of patients undergoing a radical treatment for prostate cancer such as: radical prostatectomy, radiotherapy, brachytherapy divided by the total number of patients.
Total number of cores positive for cancer | Month 24
  Total number of biopsy sample containing tumor cells at the month 24 biopsy
The rate of incontinence, erectile dysfunction, urinary symptoms | Randomisation visit, Day 7 after VTP , Month 3, Month 6, Month 9, Month 12, Month 24
  Number of patients experiencing urinary incontinence, erectile dysfunction or urinary symptoms events divided by the total number of patients.
The rate of adverse events | Screening-Month 24
  Number of patients experiencing adverse events divided by the total number of patients.
The rate of severe prostate cancer related events: cancer extension to T3, metastasis and prostate cancer related death | Screening-Month 24
  Number of patients experiencing severe prostate cancer related events: cancer extension to T3, metastasis and prostate cancer related death divided by the total number of patients.
The overall quality of life will be recorded for potential utility and descriptive studies. | Randomisation visit; Month 12; Month 24
  Results of the International Index of Erectile Function (IIEF) and International Prostate Symptoms Score (IPSS) patients questionaires.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, Professor, Principal Investigator — University College of London Hospital , United Kingdom
Locations (50):
- Dept. of Urology-University Hospitals Leuven, Leuven, Belgium
- Department of Urology-Tampere University Hospital-, Tampere, Finland
- France (17):
  - Service d'Urologie - Centre Hospitalier Universitaire d'Angers, Angers
  - CHRU Hopital Jean Minjoz, Besançon
  - Site Médipole, Cabestany
  - Polyclinique Sévigné, Cesson-Sévigné
  - Clinique d'Urologie et de Transplantation Rénale CHU Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital La Conception, Marseille
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Tenon, Paris
  - Institut Mutualiste Montsouris (IMM), Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire Lyon Sud, Pierre-Bénite
  - Polyclinique les Bleuets, Reims
  - CHU Pontchaillou, Rennes
  - Clinique Urologique Nantes, Saint-Herblain
  - Hôpital Foch, Suresnes
  - Centre Hospitalier Universitaire de Rangueil, Toulouse
- Germany (11):
  - Marien Krankenahaus GmbH, Bergisch Gladbach
  - ATURO-Gemeinschaftspraxis für Urologie und Andrologie, Berlin-Wilmersdorf
  - Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität, Dresden
  - Urologische Gemeinschaftspraxis, Emmendingen
  - Martini-Klinik am UKE Hamburg-Eppendorf Prostate Cancer Center, Hamburg
  - Vinzenz Krankenhaus - Department of Urology, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - University Hospital Schleswig-Holstein, Kiel
  - Ludwig-Maximilians-Universität München, Munich
  - Urologie 24, Nuremberg
- Italy (4):
  - Unità Operativa Urologia Lucca - c/o Azienda USL 2 - Ospedale Campo di Marte, Lucca
  - Unità di Chirurgia Urologica Mininvasiva, Roma
  - Unità Operativa Urologica di Savona, Ospedale San Paolo di Savona, Savona
  - Osp. S. Giov. Battista Molinette-Dipartimento di Discipline Medico-Chirurgiche Urologia, Torino
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Polikliniek Urologie-Catharina Ziekenhuis, Eindhoven
- Spain (8):
  - Hospital Universitari de Bellbitge-Servico de Urologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de A Coruña, A Coruña
  - Fundacio Puigvert-Department of Urology, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Department of Urology-Hospital Clinic, University of Barcelona, Barcelona
  - Hospital 12 de Octubre - Departmento de Urologia, Madrid
  - Complejo Hospitalario Regional Virgen Del Rocio-Department Urology, Seville
  - Instituto Valenciano de Oncologia, Valencia
- Dept of Urology-University Hospital-, Malmo, Sweden
- Anna-Seiler-Haus Inselspital, Bern, Switzerland
- United Kingdom (4):
  - Kings College Hospital (KCH), London
  - University College of London Hospital, London
  - Oxford John Radcliffe Hospital Trust, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data are available in case report form for each patient
Time Frame: Data available on request.

REFERENCES:
- [Result] Azzouzi AR, Vincendeau S, Barret E, Cicco A, Kleinclauss F, van der Poel HG, Stief CG, Rassweiler J, Salomon G, Solsona E, Alcaraz A, Tammela TT, Rosario DJ, Gomez-Veiga F, Ahlgren G, Benzaghou F, Gaillac B, Amzal B, Debruyne FM, Fromont G, Gratzke C, Emberton M; PCM301 Study Group. Padeliporfin vascular-targeted photodynamic therapy versus active surveillance in men with low-risk prostate cancer (CLIN1001 PCM301): an open-label, phase 3, randomised controlled trial. Lancet Oncol. 2017 Feb;18(2):181-191. doi: 10.1016/S1470-2045(16)30661-1. Epub 2016 Dec 20. PMID 28007457
- [Derived] Azzouzi AR, Barret E, Bennet J, Moore C, Taneja S, Muir G, Villers A, Coleman J, Allen C, Scherz A, Emberton M. TOOKAD(R) Soluble focal therapy: pooled analysis of three phase II studies assessing the minimally invasive ablation of localized prostate cancer. World J Urol. 2015 Jul;33(7):945-53. doi: 10.1007/s00345-015-1505-8. Epub 2015 Feb 25. PMID 25712310
- [Derived] Lebdai S, Villers A, Barret E, Nedelcu C, Bigot P, Azzouzi AR. Feasibility, safety, and efficacy of salvage radical prostatectomy after Tookad(R) Soluble focal treatment for localized prostate cancer. World J Urol. 2015 Jul;33(7):965-71. doi: 10.1007/s00345-015-1493-8. Epub 2015 Jan 23. PMID 25614256